CLINICAL TRIAL: NCT01400347
Title: Influence of Fatigue and Speed on Electromyographic Activity of Lower Extremity Muscles During Selected Weight Bearing Exercises Commonly Used for Fitness and Rehabilitation
Brief Title: Electromyography During Common Exercises Used in Rehabilitation
Status: Withdrawn | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: EMGMarko
Record Dates: First submitted 2009-11-18; First posted 2011-07-22 (Estimated); Last update posted 2021-10-22 (Actual); Status verified 2009-11

CONDITIONS: Motor Activity
Keywords: Motor activity, lower extremity, physical exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
It is generally accepted that the effectiveness of an exercise can be controlled not only by the weight or resistance applied but also by doing an exercise that would better target the desired muscle. The purpose of this study is to obtain objective information regarding selected lower extremity muscle activity during specific exercise and the influence of fatigue and speed on muscular activation.

DETAILED DESCRIPTION:
It is generally accepted that the effectiveness of an exercise can be controlled not only by the weight or resistance applied but also by doing an exercise that would better target the desired muscle. Information regarding selected lower extremity muscle activity during specific exercise and the influence of fatigue and speed on muscular activation may enhance exercise prescription for all parties involved. Specifically, selection of specific training or rehabilitation exercises may be guided by increased awareness of specific muscle activation patterns during common exercises.

Methods and Measures: Healthy subjects between 18 - 35 years old will be recruited from the community by a sample of convenience and word of mouth. Potential participants will report to the Institute for Human Performance. The potential participants will be asked to complete all documentation including informed consent, and health screening questionnaire. The qualified participants will be familiarized with the set up and specific exercises. If eligible, surface EMG recordings will be collected from the back extensors, gluteal muscles (buttocks), hamstrings (posterior thigh), quadriceps (anterior thigh), and gastrocnemius (calf) during squat and lunges exercises.

For data analysis, a within subject measures analysis will be conducted using general linear models. Specifically, we will use paired t-tests and an analysis of variance (ANOVA). When applicable, post-hoc tests will be used to uncover differences among the groups of subjects on descriptor variables such as age, height, weight, rate of perceived exertion, and maximal and sub-maximal voluntary muscle performance variables (i.e. EMG amplitude, frequency). The statistical significance level will be set at alpha = 0.05 for all analyses performed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults age 18-35

Exclusion Criteria:

* Subjects who report any significant respiratory-cardiovascular disease, which is not yet under control.
* Known orthopedic risks to strength training exercise

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We will recruit healthy, young (18-35 y.o.) subjects. Following signing the inform consent, potential participants will be given a health risk questionnaires to identify possible cardiovascular and/or orthopedic risks to strength training exercise. Answering YES to any of the questions on the PAR Q will be considered an exclusion criterion. In addition we will use a MEDICAL HISTORY QUESTIONNAIRE (included at the end of this form). Specifically, subjects who are at risk due to recent (within the last year) neuro-musculo-skeletal injury to lower extremities will be excluded from the study. Also, we will exclude subjects who reported any significant respiratory-cardiovascular disease, which is not yet under control..
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Marko, DPT, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- The Institute for Human Performance, Syracuse, New York, United States